CLINICAL TRIAL: NCT06736639
Title: Morphological Characteristics of Inferior Pole Patellar Fractures and a Finite Element Analysis Combined with a Retrospective Clinical Study of Anchor Suture and Titanium Cable Cerclage Treatment
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: JD-HG-2024-064
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Inferior Patellar Fracture; Fracture Maps; Finite Element Analysis
Keywords: Inferior Patellar Fracture; Fracture Maps; Finite Element Analysis; Retrospective Study
MeSH Terms: interventions — Suture Anchors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Anchor + titanium cable cerclage (ISB-LP): This group includes patients with inferior pole patellar fractures (IPPF) treated using anchor suture fixation combined with titanium cable cerclage. The intervention involves securing fracture fragments with anchors to provide stable fixation, reinforced by a titanium cable cerclage for additional stability. This method is intended to reduce hardware-related complications while maintaining biomechanical stability and supporting functional recovery. The outcomes for this group include operative time, postoperative knee range of motion, incidence of complications, need for secondary surgery, and functional scores such as the Bostman score.
  Interventions: Procedure: Anchor Suture with Titanium Cable Cerclage
- TBW-LP fixed (TBW-LP group): This group includes patients with inferior pole patellar fractures (IPPF) treated using Kirschner-wire tension band combined with patellar cerclage (TBW-LP group). This intervention involves the placement of Kirschner wires to create a tension band construct across the fracture site, stabilizing the fragments, with additional support provided by a cerclage wire. This method is widely used in clinical practice due to its simplicity and cost-effectiveness. The study evaluates key outcomes for this group, including operative time, knee range of motion, incidence of postoperative complications such as hardware irritation or infection, and functional recovery based on Bostman scores. This group serves as a comparison to newer techniques like anchor suture with titanium cable cerclage.
  Interventions: Procedure: Kirschner wire tension band + cerclage cable

INTERVENTIONS:
Procedure: Anchor Suture with Titanium Cable Cerclage — This intervention involves the use of **anchor suture fixation combined with titanium cable cerclage** for the treatment of inferior pole patellar fractures (IPPF). The anchor suture provides stable fixation of fracture fragments by anchoring directly into the bone, while the titanium cable cerclage offers additional reinforcement around the patella to enhance stability and minimize fragment displacement. This method is specifically designed to address the limitations of traditional Kirschner-wire tension band techniques, such as hardware irritation and infection, by using biocompatible and low-profile materials.
  Groups: Anchor + titanium cable cerclage (ISB-LP)
Procedure: Kirschner wire tension band + cerclage cable — This intervention uses **Kirschner wire tension band combined with cerclage cable** to treat inferior pole patellar fractures (IPPF). The Kirschner wires are positioned across the fracture site to form a tension band, which transforms tensile forces into compressive forces, promoting fracture stability. The cerclage cable is added to reinforce the fixation by encircling the patella, providing additional stability to comminuted or complex fractures.
  Groups: TBW-LP fixed (TBW-LP group)

SUMMARY:
The goal of this study is to compare the biomechanical stability and clinical outcomes of two treatment methods for inferior pole patellar fractures (IPPF): anchor suture with patellar cerclage and Kirschner-wire tension band combined with patellar cerclage. The study involves patients with IPPF, focusing on fracture patterns and treatment outcomes.

1. Undergo retrospective analysis of fracture patterns using fracture mapping.
2. Participate in biomechanical analysis via finite element modeling of both treatment methods.
3. Be part of a clinical comparison between two surgical treatments based on operative time, postoperative complications, and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

(1) diagnosis of IPPF confirmed by X-ray or CT, and (2) patients aged between 18 and 70 years.

Exclusion Criteria:

(1) concomitant fractures of other parts of the knee, (2) open fractures, and (3) pathological fractures.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with inferior pole patellar fractures (IPPF), confirmed through X-ray or CT imaging, and aged between 18 and 70 years. Eligible participants include individuals with isolated inferior pole patellar fractures who meet the inclusion criteria. Patients with concomitant fractures of other parts of the knee, open fractures, or pathological fractures are excluded to ensure a homogenous study population. This population represents a clinically relevant group for evaluating the outcomes of surgical interventions for IPPF.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
final knee range of motion | 6 months to 1.5 years after surgery
  The final knee range of motion is assessed to evaluate the functional recovery of patients following surgical treatment for inferior pole patellar fractures (IPPF). This measure includes the degree of flexion and extension achieved during follow-up, as documented through physical examination and patient self-reports. The range of motion is compared between the two intervention groups to determine the effectiveness of each treatment method in restoring knee functionality and mobility. Outcomes are measured and analyzed based on clinical standards and benchmarks for knee rehabilitation.
incidence of secondary surgery | 6 months to 1.5 years after surgery
  The incidence of secondary surgery is defined as the number of patients who require an additional surgical procedure related to the treatment of inferior pole patellar fractures (IPPF) within the follow-up period. This includes procedures to address complications such as hardware irritation, infection, nonunion, malunion, or mechanical failure of the initial fixation. The data will be compared between the two intervention groups to evaluate the durability and long-term effectiveness of each surgical technique. This measure provides critical insights into the need for re-intervention and overall treatment success.
postoperative complications | 6 months to 1.5 years after surgery
  Postoperative complications include any adverse events or clinical issues occurring as a result of the surgical treatment for inferior pole patellar fractures (IPPF) within the follow-up period. These complications may include, but are not limited to, hardware irritation, infection, wound dehiscence, delayed union, nonunion, or malunion. Data will be collected from medical records and follow-up visits to identify the frequency and types of complications in each intervention group. The results will be analyzed to compare the safety profiles of the anchor suture with titanium cable cerclage and the Kirschner wire tension band with cerclage cable techniques. This outcome is critical for assessing the overall safety and effectiveness of each surgical approach.

SECONDARY OUTCOMES:
operative time | 6 months to 1.5 years after surgery
  Operative time is defined as the total duration of the surgical procedure, measured from the initial incision to the completion of wound closure. This outcome measure evaluates the efficiency of the surgical intervention and provides insights into the complexity and technical demands of each technique. Operative time is compared between the two groups (anchor suture with titanium cable cerclage vs. Kirschner wire tension band with cerclage cable) to assess any significant differences in surgical duration. This metric is particularly relevant in evaluating the practicality and feasibility of each intervention in clinical practice.
functional recovery | 6 months to 1.5 years after surgery
  Functional recovery is evaluated using validated scoring systems, such as the Bostman score, to assess the restoration of knee function following surgical treatment for inferior pole patellar fractures (IPPF). This measure includes parameters such as pain levels, range of motion, ability to perform daily activities, and overall patient satisfaction. Data will be collected during follow-up visits to determine the extent of functional improvement and to compare outcomes between the two intervention groups (anchor suture with titanium cable cerclage vs. Kirschner wire tension band with cerclage cable). This outcome provides critical insights into the effectiveness of each surgical technique in achieving optimal rehabilitation and long-term knee function.

CONTACTS AND LOCATIONS:
Locations (1):
- The medical record system and imaging system of the Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Hu Z, Sun C, Heng H, Li J, Chen H, Chen F, Su P, Wang D. Morphological Characteristics of Inferior Pole Patellar Fractures and a Finite-Element Analysis Combined With a Retrospective Clinical Study of Anchor Suture and Titanium Cable Cerclage Treatment. Orthop Surg. 2025 Apr;17(4):1045-1056. doi: 10.1111/os.14351. Epub 2025 Jan 22. PMID 39844589